CLINICAL TRIAL: NCT05447676
Title: Effects of 4-AP on Functional Recovery After Spinal Cord Injury
Brief Title: Effects of 4-AP on Functional SCI Recovery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Monica Perez, Chair, Arms and Hands, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00215984; R35NS122336 (NIH)
Record Dates: First submitted 2022-06-20; First posted 2022-07-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injury
Keywords: SCI; Neural control; 4-AP; Walking; Neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries | interventions — 4-Aminopyridine; Exercise

STUDY DESIGN:
Intervention Model Description: Arm 1 and 2 will be studied with randomized crossover design; Participants for Arm 3 will be recruited after finishing the sessions for Arms 1 and 2. Participants who were finished the Arms 1 and 2 study procedures can also participate in Arm 3 study procedures.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not know if they receive 4-AP or placebo over the course of the study and the investigators are also blinded except for PI (Dr. Monica Perez).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dalfampridine (4-AP)+STDP+training (Active Comparator): The effects of the functional recovery of the lower-limb muscles will be determined after 10 sessions of 4-AP, STDP stimulation and training.
  Interventions: Drug: Dalfampridine; Other: STDP stimulation; Behavioral: Exercise training
- Placebo+STDP+training (Placebo Comparator): The effects of the functional recovery of the lower-limb muscles will be determined after 10 sessions of placebo drug, STDP stimulation and training.
  Interventions: Other: Placebo drug; Other: STDP stimulation; Behavioral: Exercise training
- Dalfampridine (4-AP)+STDP+training for extended sessions (Experimental): The long-term effects of the functional recovery of the lower-limb muscles will be determined after 40 sessions of 4-AP, STDP stimulation and training.
  Interventions: Drug: Dalfampridine; Other: STDP stimulation; Behavioral: Exercise training

INTERVENTIONS:
Drug: Dalfampridine — The study drug (4-AP) will be administered as a 10 mg dose.
  Other Names: 4-AP
  Arms: Dalfampridine (4-AP)+STDP+training; Dalfampridine (4-AP)+STDP+training for extended sessions
Other: Placebo drug — The pharmacy will also provide a placebo drug that looks identical to 4-AP to verify participants and therapists do not know who is receiving the drug and who is receiving the placebo.
  Arms: Placebo+STDP+training
Other: STDP stimulation — Paired stimulation will be given to the spinal cord and to peripheral nerves so that the signals are received at the spinal cord at a specific interval.
  Other Names: spike timing dependent plasticity
Behavioral: Exercise training — Lower-limb exercises will involve over-ground walking, treadmill, walking and stair climbing training.

SUMMARY:
The purpose of this study is to test a strategy to potentiate functional recovery of lower limb motor function in individuals with spinal cord injury (SCI). The FDA approved drug, Dalfampridine (4-AP). 4-AP will be used in combination of Spike-timing-dependent plasticity (STDP) stimulation and STDP stimulation with limb training.

DETAILED DESCRIPTION:
Currently, research has shown that 4-AP has a positive effect on sensory and motor function rehabilitation in humans with chronic SCI in addition to decreasing recorded spasticity, increased sensation, and decreased pain. Utilizing limb training to promote recovery of motor function is enhanced by eliciting STDP in the limbs. An important strength of this aim is the combination of training and STDP, which aims at enhancing the beneficial effects of motor training by promoting plasticity in the corticospinal pathway. We hypothesize that introducing 4-AP into the STDP stimulation and STDP stimulation with lower-limb training will further improve motor function rehabilitation in patients with chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between ages 18-85 years
* SCI at least 4 weeks post injury
* Spinal Cord injury at or above L2
* ASIA A,B,C, or D, complete or incomplete
* Possess the following abilities
* The ability to perform a small visible contraction with dorsiflexion and hip flexor muscles

Exclusion Criteria:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any history of renal impairment
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without history of seizure, and without anticonvulsant medication
* History of seizures or epilepsy
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold (see appendix 2)
* Pregnant females
* If a women of child bearing age is unsure of the pregnancy, and does not want to take the pregnancy test Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated disk
* Metal plate in skull
* Individuals with scalp shrapnel, cochlear implants, or aneurysm clips
* Individuals taking Bupropion, Dolutegravir, Lacosamide, Trilaciclib, or PR Interval prolonging drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in TMEPs | TMEPs measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training and Placebo+STDP+training groups. TMEPs measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  Electrical stimulation will be performed placing the cathode on the upper thoracic between the spinal processes between T3 and T4 vertebrae and the anode at ~10 cm above
Change in MVC | MVC measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training and Placebo+STDP+training groups. MVC measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  Individuals will perform a maximum voluntary contraction (MVC) of each targeted muscle (quadriceps femoris, tibialis anterior or soleus) through surface electrodes secured to the skin over the belly of each muscle.

SECONDARY OUTCOMES:
Change in MEPs | MEPs measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training and Placebo+STDP+training groups. MEPs measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  Transcranial magnetic stimuli (TMS) will be delivered to the optimal scalp position for activation of quadriceps femoris and tibialis anterior muscles. The optimal scalp position will be determined by moving the coil in small steps along the hand/arm/leg representation of the primary motor cortex to find the region where the largest MEP can be evoked with the minimum intensity in the targeted muscles.
Change in 10-meter walk test | 10-m walk measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training and Placebo+STDP+training groups. 10-m walk measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  We will use the 10-meter walk test to quantify walking speed in meters per second. The same percentage of body-weight support will be used during pre- and post-assessments. Less time to walk 10-meter indicates better outcome.
Change in 6-minute walk test | 6-min walk measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training & Placebo+STDP+training groups. 6-min walk measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  We will measure the distance walked over 6 minutes. The same percentage of body-weight support will be used as in 10-meter walk test. The longer distance walked during 6 minutes indicates better outcome.
Change in International Standards for Neurological Classification of Spinal Cord Injury exam | Scores measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training and Placebo+STDP+training groups. Scores measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  Motor part of the exam is completed through the testing of key muscle functions corresponding to 10 myotomes (C5-T1 and L2-S1) for right and left side separately. The strength of each muscle function is graded on a six-point scale ranging from 0 meaning complete paralysis to 5 meaning full strength. The total motor score is sum of all motor scores range from 0-100. Sensory part of the exam is completed through the testing of a key point in each of the 28 dermatomes (from C2 to S4-5) on the right and left sides of the body. At each of these key points, two aspects of sensation are examined: light touch and pin prick. Appreciation of light touch and pin prick sensation at each of the key points is separately scored on a three-point scale; 0-absent, 1-altered, and 2-normal or intact. 56 is the maximum score for both light touch and pin prick and the total sensory score ranges from 0 to 112. Higher scores represent better outcome for motor and sensory scores.
Change in surveys on ambulation, basic mobility, bowel and bladder management difficulties | SCI-QOL measured at baseline and 3 weeks (10 sessions) for Dalfampridine+STDP+training & Placebo+STDP+training groups. SCI-QOL measured at baseline, 6 weeks (20 sessions), and 12 weeks (40 sessions) for extended sessions group.
  The name of the questionnaire is Spinal Cord Injury Quality of Life (SCI-QOL) and we used four subdomains: ambulation, self-care, bowel management difficulties, and bladder management difficulties. Scores on all subdomains of SCI-QOL use a standardized T metric, with a mean of 50 and a standard deviation of 10. Ambulation and basic mobility subdomains assess the ability to engage in walking activities in different locations that vary based on speed, time and condition and the ability to manage stairs under different conditions. Bowel management difficulties subdomain measures an ability to carry out a bowel program; concerns about incontinence and bowel accidents; and the impact of bowel management on everyday living. Bladder management difficulties subdomain measures ability to carry out a bladder program; worry about bladder accidents; concerns about implementing one's bladder program; and impact on everyday living. Higher scores on all subdomains represent better outcome.
Change in morphological characterization of corticospinal and reticulospinal pathways in MRI | MRI measured at baseline and 12 weeks (40 sessions) for Dalfampridine+STDP+training for extended sessions group.
  In order to identify descending motor tract, brainstem and C2 cervical spinal cord images will be acquired on a MAGNETOM Prisma 3T system using a 64-channel birdcage head/neck coil. To quantify the effect of atrophy in oblique directions, we will measure the radius from the cord shape center of mass to its border, R(α), for angles α over the whole circle with an angular resolution of 6°. Mean measures of all 5 axial slices will be used for statistical from nerve roots, noise, and other confounding effects.

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PT, PhD, Principal Investigator — Shirley Ryan Ability Lab
Locations (1):
- Shirley Ryan Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No